CLINICAL TRIAL: NCT02091687
Title: Longitudinal Outcomes in Pediatric rTMS and CIT
Acronym: Longitudinal
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1401S47261
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Congenital Hemiparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Track behavioral and qualitative longitudinal outcomes in children with hemiparesis who previously participated in a randomized, controlled trial (RCT) of intensive therapy combined with repetitive Transcranial Magnetic Stimulation (rTMS)

DETAILED DESCRIPTION:
This longitudinal study will evaluate the subjective and behavioral outcomes of a previous randomized controlled study (RCT) rTMS/CIT (Pediatric Hemiparesis: Synergistic Treatment using rTMS and CIT (NIH Grant Number: 1RC1HD063838-01; PI: Dr. James Carey). The previous rTMS/CIT study evaluated the safety and efficacy of 5 treatments of 6-Hz primed low-frequency rTMS applied to the non-stroke hemisphere combined with constraint induced therapy (CIT) to promote recovery of the paretic hand in children and adolescents. CIT has shown improved behavioral outcomes as well as cortical reorganization in representation of the affected limb. The previous RCT was a rTMS-Sham/CIT study design (real rTMS n=10 and sham rTMS n=9).

Our research question, 'What is the medical status and perception of previous participants concerning their involvement in an intensive rTMS/CIT RCT specific to symptom monitoring, the TMS experience, and their current functional status'.

ELIGIBILITY:
Inclusion Criteria:

* Previous participants in a RCT on rTMS/CIT.

Exclusion Criteria:

* Participants who do not wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previous participants in a randomized controlled study (RCT) rTMS/CIT (Pediatric Hemiparesis: Synergistic Treatment using rTMS and CIT (NIH Grant Number: 1RC1HD063838-01; PI: Dr. James Carey)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
TMS Symptom Checklist | Adminstered at testing session, 2-4 years after intervention.
  This checklist assists in monitoring children who have had TMS for side effects.

SECONDARY OUTCOMES:
Assisting Hand Assessment | at testing session, 2-4 years after intervention.
  This assessment evaluates how well a child can use his/her hands during every day two handed activities.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette T Gillick, PhD, MSPT, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Rich TL, Menk J, Krach LE, Feyma T, Gillick BT. Repetitive Transcranial Magnetic Stimulation/Behavioral Intervention Clinical Trial: Long-Term Follow-Up of Outcomes in Congenital Hemiparesis. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):598-605. doi: 10.1089/cap.2015.0157. Epub 2016 Feb 23. PMID 26905272
- [Background] Rich T, Cassidy J, Menk J, Van Heest A, Krach L, Carey J, Gillick BT. Stability of stereognosis after pediatric repetitive transcranial magnetic stimulation and constraint-induced movement therapy clinical trial. Dev Neurorehabil. 2017 Apr;20(3):169-172. doi: 10.3109/17518423.2016.1139008. Epub 2016 Mar 17. PMID 26985568